CLINICAL TRIAL: NCT01786564
Title: Home Sleep and Circadian Phase: Mediators of Diabetes Risk
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Kristen Knutson, Associate Professor, Northwestern University
Other Study IDs: STU00204605
Record Dates: First submitted 2013-02-04; First posted 2013-02-08 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Sleep Deprivation; Diabetes; Circadian Dysregulation
Keywords: diabetes; sleep
MeSH Terms: conditions — Sleep Deprivation; Diabetes Mellitus; Chronobiology Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to determine if deficient sleep and/or disruption with the body's internal clock ("circadian rhythms") are associated with diabetes risk. This study is being done to look at the possible relationships between sleep and risk of diabetes by examining sleep in the home and diabetes risk in the laboratory.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 21-50 years
2. BMI <40 kg/m2.
3. No major illness.
4. No history of psychiatric, endocrine, cardiac or sleep disorders,
5. Premenopausal, non-pregnant women.
6. Those with dyslipidemia and hypertension will be included if these conditions are controlled by a stable treatment, such as lipid-lowering or antihypertensive medications (except beta blockers).

Exclusion criteria include:

1. Persons with diabetes.
2. Persons with diagnosed sleep disorders or apnea-hypopnea index>15.
3. History of cardiovascular event or disease (excluding controlled hypertension).
4. Major psychiatric disorder or other major illness.
5. Persons taking medications, including but not limited to antidepressants and hypnotics (but excluding lipid-lowering drugs and anti-hypertensive medications as mentioned above).
6. Persons regularly taking medication that affects melatonin such as beta blockers and exogenous melatonin.
7. Anyone who tests positive for common drugs of abuse.
8. People with color blindness.
9. People who have had Lasik eye surgery.
10. People who work night shifts.
11. Participants who travel across multiple time zones will be studied only after they have remained in the Central Time Zone (or Indiana) for one month prior to the study.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study will recruit a total of 100 African Americans (AA) and 100 non-Hispanic whites (WH) with equal numbers of men and women in each group completing the entire study. Ages will be 21-50 years and body mass indices (BMI) will be <40 kg/m2.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2011-12-06 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Knuston, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 120 participants enrolled in the study, 56 were eligible, continued in the study and provided some data.
Groups:
- Study Sample: This is a cross-sectional study so there is only one group.
Period: Overall Study
Arm/Group | Study Sample
Started | 120
Completed | 56
Not Completed | 64
Not completed — Lost to Follow-up | 47
Not completed — Ineligible | 17

BASELINE CHARACTERISTICS:
Arm/Group | Study Sample
Number analyzed (Participants) | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 56
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 27
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 56
Body Mass Index (BMI), kg/m2 [Mean (Standard Deviation); unit: kg/m2] | 27.7 (5.3)
Habitual Sleep Duration (hours) [Mean (Standard Deviation); unit: minutes] — Population: Three participants did not have valid actigraphy data so habitual sleep measures could not be calculated. Thus only 53 participants have habitual sleep measures.
  minutes
    number analyzed (Participants) | 53
    (all) | 402 (39)
Habitual sleep efficiency (% of sleep period sleeping) [Mean (Standard Deviation); unit: percentage] — Population: Three participants did not have valid actigraphy data so habitual sleep measures could not be calculated. Thus only 53 participants have habitual sleep measures.
  percentage
    number analyzed (Participants) | 53
    (all) | 90.8 (3.5)
Habitual sleep start time (clock time) [Mean (Standard Deviation); unit: Hours after midnight] — Population: Three participants did not have valid actigraphy data so habitual sleep measures could not be calculated. Thus only 53 participants have habitual sleep measures.
  Hours after midnight
    number analyzed (Participants) | 53
    (all) | 0.27 (1.51)
Duration of Stage 2 sleep (minutes) [Mean (Standard Deviation); unit: Minutes] — Population: Five participants did not have a valid PSG recording. Thus only 51 participants have sleep stage data.
  Minutes
    number analyzed (Participants) | 51
    (all) | 190.6 (77.4)
Duration of Stage 3 sleep (minutes) [Mean (Standard Deviation); unit: Minutes] — Population: Five participants did not have a valid PSG recording. Thus only 51 participants have sleep stage data.
  Minutes
    number analyzed (Participants) | 51
    (all) | 68.4 (30.7)
Duration of Rapid Eye Movement (REM) sleep (minutes) [Mean (Standard Deviation); unit: Minutes] — Population: Five participants did not have a valid PSG recording. Thus only 51 participants have sleep stage data.
  Minutes
    number analyzed (Participants) | 51
    (all) | 96.5 (49.1)
Fasting glucose levels (mg/dl) [Mean (Standard Deviation); unit: mg/dl] — Population: 2 participants were missing valid fasting blood samples so only 54 have a HOMA measure.
  mg/dl
    number analyzed (Participants) | 54
    (all) | 86.8 (6.3)
Estimated Insulin Resistance (HOMA index method) [Mean (Standard Deviation); unit: None (Index)] — Population: 2 participants were missing valid fasting blood samples so only 54 participants have HOMA estimated.
  None (Index)
    number analyzed (Participants) | 54
    (all) | 1.75 (1.82)
Oral Disposition Index at 30 minutes [Mean (Standard Deviation); unit: None (Index)] — Population: 3 participants were missing some blood samples so the oral disposition index could not be calculated in these 3 participants. Thus, only 53 participants have this measure.
  None (Index)
    number analyzed (Participants) | 53
    (all) | 11.5 (12.7)

OUTCOME MEASURES:

1. Primary Outcome: Oral Disposition Index
Description: The oral disposition index is based on the glucose and insulin levels during the first 30 minutes of a frequently sampled 5-hour oral glucose tolerance test. It reflects the combination of insulin sensitivity and insulin release in response to the glucose challenge. Higher values suggest a greater response.
Time Frame: baseline
Population: Three participants did not have adequate glucose and/or insulin values to calculate the disposition index.
Measure: Mean (Standard Deviation); unit: None (Index)
Arm/Group | Study Sample
Number analyzed (Participants) | 53
None (Index) | 11.5 (12.7)
Statistical Analysis 1: Comparison: Study Sample; The cross-sectional association between habitual sleep duration and oral disposition index was analyzed; Test type: Other — This is cross-sectional analysis in a single group; p = .13, Regression, Linear — Unadjusted association. A priori p value of .05 was selected for statistical significance; Regression Coefficient = -.075, 95% CI 2-sided [-.173 to .023]
Statistical Analysis 2: Comparison: Study Sample; The cross-sectional association between habitual sleep quality (sleep percentage) and oral disposition index was analyzed; Test type: Other — This is cross-sectional analysis; p = .83, Regression, Linear — Unadjusted association. P value of .05 was selected a priori as statistical significance; Unadjusted; Regression Coefficient = 0.12, 95% CI 2-sided [-0.95 to 1.19]
Statistical Analysis 3: Comparison: Study Sample; The cross-sectional association between amount of Stage 3 sleep and oral disposition index was analyzed; Test type: Other — This is cross-sectional analysis in a single group; p = .39, Regression, Linear — Unadjusted association. A priori p value of .05 was selected for statistical significance; Unadjusted; Regression Coefficient = -.05, 95% CI 2-sided [-.166 to 0.66]
Statistical Analysis 4: Comparison: Study Sample; The cross-sectional association between amount of REM sleep and oral disposition index was analyzed; Test type: Other — Unadjusted association. P value of .05 was selected a priori as statistical significance; p = .11, Regression, Linear — Unadjusted association. P value of .05 was selected a priori as statistical significance; Unadjusted association; Regression Coefficient = -.058, 95% CI 2-sided [-.129 to .014]

ADVERSE EVENTS:
Time Frame: During study participation, approximately 2 weeks.
Description: Definitions do not differ.
Arm/Group | Study Sample
All-Cause Mortality (participants affected / at risk) | 0/56
Serious Adverse Events (participants affected / at risk) | 0/56
Other Adverse Events (participants affected / at risk) | 0/56

LIMITATIONS AND CAVEATS:
Study sample was lower than anticipated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-05-24): https://cdn.clinicaltrials.gov/large-docs/64/NCT01786564/Prot_SAP_ICF_001.pdf